CLINICAL TRIAL: NCT03540563
Title: Prospective Study Evaluating ctDNA as a Biomarker for Treatment Response in Head and Neck Squamous Cell Carcinoma'
Brief Title: ctDNA as a Biomarker for Treatment Response in HNSCC
Acronym: PECAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N18PCN
Record Dates: First submitted 2018-03-14; First posted 2018-05-30 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: ctDNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood draw (Other): Blood and saliva specimens will be taken for ctDNA analysis at baseline, weekly during treatment and at 2 weeks after treatment. During follow up both blood and saliva will be obtained in combination with a CT/MRI scan on the same day at 3 months, 6 months, 1 year and 2 years after treatment.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood will be drawn to assess ctDNA

SUMMARY:
Tumours continually shed DNA into the circulation, where it can be accessed. This circulating tumour DNA (ctDNA) directly reflects tumour burden and has great potential to be a sensitive biomarker for treatment recurrence. These "liquid biopsies" could give a more real-time picture of the genomic status and evolution of a tumour and can be easily assessed for measurement of different biomarkers. However, in head and neck squamous cell carcinoma (HNSCC) patients treated with primary curative radiotherapy, data regarding ctDNA kinetics and its correlation with outcome are scarce. A new or additional tool for response evaluation next to or instead of conventional imaging after treatment would be beneficial to detect recurrences in an earlier stage, thereby increasing the chances of success of salvage therapy. More importantly, an early response parameter during treatment could help to identify patients that have a good treatment response and might benefit from treatment adaptation. With this study, we aim to reveal ctDNA as an effective tool for future dose (de)-escalation trials in HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Stage II-IV carcinoma of the larynx, hypopharynx, oral cavity or HPV negative oropharynx or stage II-III HPV positive oropharyngeal carcinoma, histologically confirmed according to the American Joint Committee on Cancer (AJCC) staging manual 8th edition
* Indication for primary curative radiotherapy with or without concurrent radio sensitizer
* WHO performance status 0-2
* Signed written IC

Exclusion Criteria:

* Metastatic disease
* Radiotherapy with palliative intent
* Diagnosis of any other malignancy within 5 years prior to start of treatment except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, or low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (e.g. surgery, radiation or castration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The number of patients in which ctDNA measurement (in amplifiable copies per millilitre blood and saliva) accurately predicts treatment outcome within 2 years after treatment, in terms of FFP. | 2 years
  ctDNA biomarker

SECONDARY OUTCOMES:
CtDNA kinetics (clearance time, drop below a certain level, complete absence, etc.) during radiotherapy as a predictor for disease recurrence within 2 years after treatment, in terms of FFP. | 2 years
  ctDNA biomarker
Levels of ctDNA at the time of corresponding conventional imaging in relation to disease occurrence. | 3 years
  ctDNA biomarker
The number of traceable mutations found in blood / saliva in comparison with mutations found in tissue biopsies. | 3 years
  ctDNA biomarker
The tumours' genomic status and epigenetic evolution over time under pressure of radiotherapy, in terms of number of different detectable mutations at all specified time points. | 3 years
  ctDNA biomarker
Levels of ctDNA in blood compared to saliva at the same time points. | At study completion, after 3 years
  ctDNA biomarker
Levels of ctDNA before treatment compared to other clinical/biological parameters in the prediction of treatment response. | 3 years
  ctDNA biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Abrahim Al-Mamgani, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Patients sign for participation in this study and not for use in other studies